CLINICAL TRIAL: NCT06315270
Title: To Explore the Feasibility of Dynamic Changes of TCR Diversity in Peripheral Blood in Monitoring Recurrence and Evaluating Prognosis of Epithelial Ovarian Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 24K040-001
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-01

CONDITIONS: Epithelial Ovarian Cancer; Stage III Ovarian Cancer; Stage IV Ovarian Cancer
Keywords: TCR; Immunological monitoring
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project proposes to elucidate the functional impact of T cells in cancer progression and treatment through a comprehensive TCR profiling study and a longitudinal cohort study in patients with advanced epithelial ovarian cancer. Our findings aim to provide clinical insights for monitoring treatment response in a non-invasive way and demonstrate the association of TCR diversity with clinical outcomes and the potential role of TCR profiling in cancer prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with advanced EOC, 18-75 years of age: including patients with preoperative assessment of stage III-IV EOC, who underwent initial tumour cytoreduction and 6-8 courses of postoperative chemotherapy with paclitaxel + carboplatin/docetaxel + carboplatin;
* Eastern Cooperative Oncology Group (ECOG) physical strength status (PS) score of 0 or 1;
* Cooperation in the treatment process by providing clinicopathological data and imaging data required for the study process;
* Cooperate with follow-up visits and collection of node blood for clinical efficacy assessment, and agree to use the test data for subsequent research and product development.
* The initial and follow-up treatment processes are in accordance with NCCN guidelines;

Exclusion Criteria:

* Neoadjuvant chemotherapy patients;
* Splenectomy patients;
* Patients with contraindications to radiotherapy;
* Any other patients who, in the judgement of the investigator, may have poor compliance with the procedures and requirements of the study;
* Unacceptable or unavailable means of assessing specified efficacy such as imaging;
* Vaccination within 2 months; antibiotics for infection within 2 weeks; history of blood transfusion within 2 weeks;
* Long-term use of recombinant human erythropoietin, recombinant human interleukin, Ricodin tablets and other drugs affecting the composition of blood cells;
* Severe organ dysfunction;
* Infectious diseases such as immunodeficiency syndrome, active tuberculosis, HIV infection, and other infectious diseases not suitable for participation;
* Pre-cancerous diseases of the blood, such as myelodysplastic syndromes;
* Have received immunosuppressive therapy within 2 weeks;
* Suffering from blood clotting disorders.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynaecological cancers
Study Population: advanced EOC
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2029-03-20 (Estimated); Study Completion 2029-03-20 (Estimated)

PRIMARY OUTCOMES:
Analysis of TCR genealogy data | 5 years
  1. Analysis of TCRα and TCRβ profile profiles in advanced EOC patients before initial treatment;
  2. Analysis of differences in diversity of TCRα and TCRβ profiles in advanced EOC patients before treatment, after completion of treatment and at relapse;
  3. Analysis of longitudinal TCR profiles revealing the stability and individual specificity of the immune profiles;
  4. correlation of TCRα and TCRβ profiling diversity with levels of tumour markers (ca125, ca199, CEA, HE-4) and imaging findings under continuous monitoring to explore their value in monitoring tumour treatment response
  5. Differential analysis of dynamic changes in TCRα profile and TCRβ profile in correlation with patients' clinical outcomes

IPD SHARING:
Plan to Share IPD: No